CLINICAL TRIAL: NCT05239741
Title: A Phase 3 Study of Pembrolizumab (MK-3475) Versus Chemotherapy in Chinese Participants With Stage IV Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Colorectal Cancer (MK-3475-C66)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Chemotherapy in Chinese Participants With Stage IV Colorectal Cancer (MK-3475-C66)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-C66; MK-3475-C66 (Other: MSD)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 treatments (approximately 2 years).
  Interventions: Biological: Pembrolizumab
- Standard of Care Chemotherapy (Active Comparator): Participants receive 1 of 6 possible standard chemotherapy regimens at the discretion of the investigator: (1) mFOLFOX6; (2) mFOLFOX6+bevacizumab 5 mg/kg IV on Day 1 of each 14-day cycle (Q2W); (3) mFOLFOX6+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly Q2W; (4) FOLFIRI; (5) FOLFIRI+bevacizumab 5 mg/kg IV on Day 1 Q2W; OR (6) FOLFIRI+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly Q2W. Participants with documented disease progression following chemotherapy can receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 treatments (approximately 2 years).
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-fluorouracil; Drug: Irinotecan; Biological: Bevacizumab; Biological: Cetuximab

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: Oxaliplatin — 85 mg/m^2 given as an intravenous infusion (IV) on Day 1 in each 14-day cycle (Q2W) as part of the mFOLFOX6 regimen
  Arms: Standard of Care Chemotherapy
Drug: Leucovorin — 400 mg/m^2 given as an IV on Day 1 Q2W as part of the mFOLFOX6 and FOLFIRI regimens
  Arms: Standard of Care Chemotherapy
Drug: 5-fluorouracil — 400 mg/m^2 given as an IV bolus on Day 1 and then 1200 mg/m^2/day IV over 2 days for a total dose of 2400 mg/m^2 Q2W as part of the mFOLFOX6 and FOLFIRI regimens
  Other Names: 5-FU
  Arms: Standard of Care Chemotherapy
Drug: Irinotecan — 180 mg/m^2 IV on Day 1 Q2W as part of the FOLFIRI regimen
  Arms: Standard of Care Chemotherapy
Biological: Bevacizumab — IV infusion
  Arms: Standard of Care Chemotherapy
Biological: Cetuximab — IV infusion
  Arms: Standard of Care Chemotherapy

SUMMARY:
In this study, Chinese participants with MSI-H or dMMR advanced colorectal cancer will be assigned to receive either pembrolizumab or the Investigator's choice of 1 of 6 standard of care (SOC) chemotherapy regimens for treatment. There is no hypothesis testing for this study.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Has a histologically confirmed diagnosis of colorectal adenocarcinoma that is at stage IV (as defined by American Joint Committee on Cancer eighth edition) [National Comprehensive Cancer Network 2018]
* Has centrally confirmed Microsatellite Instability-High/Mismatch Repair Deficient (MSI-H/dMMR) status
* Has centrally confirmed RAS and BRAF mutation status
* A woman of child-bearing potential (WOCBP) must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours for urine or within 72 hours for serum before the first dose of study intervention.
* Has measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by the local site investigator/radiology
* Must provide an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 3 days before randomization
* Has a life expectancy of at least 3 months
* Has received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable hepatitis B virus (HBV) viral load prior to randomization if hepatitis B surface antigen (HBsAg) positive
* Has an undetectable Hepatitis C Virus (HCV) viral load if HCV infected
* Has well controlled Human Immunodeficiency Virus (HIV) on antiretroviral therapy (ART) if HIV infected

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* Has received prior systemic therapy for stage IV colorectal cancer (CRC). Participants may have received prior adjuvant/neoadjuvant chemotherapy for CRC as long as it was completed at least 6 months prior to randomization
* Has undergone major operation within 4 weeks of randomization or has not adequately recovered from major surgery or has ongoing surgical complications
* Has received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137])
* Has received prior radiotherapy within 2 weeks of start of study intervention or has radiation-related toxicities, requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years, with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy (eg, tuberculosis, known viral or bacterial infection)
* Has HIV-infection with a history of Kaposi's sarcoma or Multicentric Castleman's Disease
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2028-09-19 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) For All Participants | Up to approximately 77 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by BICR will be reported for all participants.
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) For RAS Wild-type Participants | Up to approximately 77 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by BICR will be reported for RAS wild-type participants .

SECONDARY OUTCOMES:
Overall Survival (OS) For All Participants | Up to approximately 77 months
  OS is defined as the time from randomization to death due to any cause. The OS will be reported for all participants.
Overall Survival (OS) For RAS Wild-type Participants | Up to approximately 77 months
  OS is defined as the time from randomization to death due to any cause. The OS will be reported for RAS wild-type participants.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) For All Participants | Up to approximately 77 months
  ORR is defined as the percentage of participants who have a best response of confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage for all participants who experience CR or PR as assessed by BICR will be presented.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) For RAS Wild-type Participants | Up to approximately 77 months
  ORR is defined as the percentage of participants who have a best response of confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage for RAS wild-type participants who experience CR or PR as assessed by BICR will be presented.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 77 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 77 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (32):
- China (32):
  - Beijing Cancer hospital-Digestive Oncology ( Site 0001), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-Medical Oncology ( Site 0011), Beijing, Beijing Municipality
  - Tianjin Medical University Cancer Institute and Hospital-Gastric oncology ( Site 0019), Tianjin, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University ( Site 0051), Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital-Medical Oncology ( Site 0012), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0009), Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center ( Site 0047), Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital ( Site 0035), Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University ( Site 0014), Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University-Oncology ( Site 0048), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College ( Site 0036), Shantou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 0039), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 0007), Harbin, Heilongjiang
  - Henan Cancer Hospital-henan cancer hospital ( Site 0015), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology-oncology ( Site 0018), Wuhan, Hubei
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 0008), Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University ( Site 0031), Changsha, Hunan
  - The Affiliated Jiangyin Hospital of Southeast University Medical College ( Site 0037), Jiangyin, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Oncology ( Site 0002), Nanjing, Jiangsu
  - The first affiliated hospital of China medical university ( Site 0043), Shemyang, Liaoning
  - Tangdu Hospital of Fourth Military Medical University of Chi-General Surgery ( Site 0045), Xi'an, Shaanxi
  - Jinan Central Hospital-oncology department ( Site 0021), Jinan, Shandong
  - Shandong Cancer Hospital ( Site 0041), Jinan, Shandong
  - Fudan University Shanghai Cancer Center-Oncology ( Site 0046), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 0022), Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital ( Site 0024), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 0032), Taiyuan, Shanxi
  - Sichuan Cancer Hospital. ( Site 0050), Chengdu, Sichuan
  - West China Hospital, Sichuan University ( Site 0044), Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University ( Site 0049), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital-Colorectal surgery ( Site 0006), Kunming, Yunnan
  - Zhejiang Cancer Hospital-oncology-abdominal neoplasms ( Site 0028), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com